CLINICAL TRIAL: NCT02500511
Title: Duration of Protection Based on Persistent Antibody Titers 12-24 Months After Vaccination: Follow Up to Phase 2 Study of Meningococcal Serogroups A, C, Y & W-135 Polysaccharide Diphtheria Toxoid Conjugate Vaccine (NmVac4-A/C/Y/W-135-DT)
Brief Title: Persistence of Protective Antibody Titers 12-24 Months After NmVac4-A/C/Y/W-135-DT Vaccination: Follow Up Study
Status: Completed | Type: Observational
Sponsor: JN-International Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: JN-NM-002E1
Record Dates: First submitted 2015-07-14; First posted 2015-07-16 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2015-07

CONDITIONS: Meningococcal Meningitis; Meningococcal Infections
MeSH Terms: conditions — Meningitis, Meningococcal; Meningococcal Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Serum samples used for antibody assays.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: NmVac4-A/C/Y/W-135-DT™ — no intervention in this study, received test vaccine in trial JN-NM-002
  Other Names: meningococcal meningitis conjugate vaccine quadrivalent

SUMMARY:
To determine the persistence of protective antibody levels for subjects who seroconverted after vaccination with NmVac4-A/C/Y/W-135-DT™

Participants in trial # JN-NM-002, who seroconverted for serogroups A and C will be contacted and asked to provide a blood sample at 12-24 months after vaccination with NmVac4-A/C/Y/W-135-DT.

Serum Bactericidal Assays will be performed to evaluated duration of protective antibody titer for NmVac4-A/C/Y/W-135-DT for all four serogroups. To determine if subjects who seroconverted with lower titers retain protective levels of antibody (titer ≥:8) at 12-24 months after vaccination.

DETAILED DESCRIPTION:
The purpose of this study is to collect serum samples to evaluate duration of protection for NmVac4-A/C/Y/W-135-DT, based on titers determined by Serum Bactericidal Assay with human complement (hSBA). This assay is used to evaluate immunogenicity of meningococcal vaccines, as a surrogate for efficacy. A titer ≥ 1:8 is considered protective.

Objectives are to evaluate duration of protective antibody titer for NmVac4-A/C/Y/W-135-DT for all four serogroups, and determine if subjects with lower titers, but ≥:8 retain protective levels of antibody at 12-24 months.

Participants in trial # JN-NM-002, who seroconverted for serogroups A and C will be contacted and asked to provide a blood sample at 12-24 months after vaccination with NmVac4-A/C/Y/W-135-DT™.

Serum Bactericidal Assays will be performed to evaluated persistence of protective antibody titer for NmVac4-A/C/Y/W-135-DT for all four serogroups, to determine if subjects who seroconverted with lower titers retain protective levels of antibody (titer ≥:8) at 12-24 months after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent
* Participant in trial JN-NM-002
* Seroconverted in trial JN-NM-002 for both serogroups A and C

Exclusion Criteria:

* Chronic medication use or medical history that, in the opinion of the Investigator, may impact the quality of the sample or safety of the subject

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects who seroconverted for serogroups A and C after vaccination with NmVac4-A/C/Y/W-135-DT in study JN-NM-001
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-06; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Antibody titer | 12-24 months after vaccination in study JN-NM-002

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Yataco, MD, Principal Investigator — IRC Clinics
Locations (1):
- IRC Clinics, Towson, Maryland, United States